CLINICAL TRIAL: NCT04817969
Title: Persona® Ti-Nidium® Personalized Total Knee System A Post-Market Clinical Follow-up Study to Provide Safety, Performance and Clinical Benefits Data Using the Persona Ti-Nidium Total Knee System and Instrumentation
Brief Title: Persona Ti-Nidium Post-Market Clinical Follow-up
Acronym: TKA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMG2020-05K
Record Dates: First submitted 2021-03-23; First posted 2021-03-26 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Knee Pain Chronic; Osteoarthritis; Rheumatoid Arthritis; Traumatic Arthritis; Polyarthritis; Varus Deformity; Valgus Deformity; Flexion Deformity of the Knee; Avascular Necrosis; Patellofemoral Osteoarthritis
Keywords: Osteoarthritis; Rheumatoid Arthritis; Total Knee Arthroplasty
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Arthritis; Osteonecrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Persona Ti-Nidium (Other): Primary total knee arthroplasty subjects that receive the Zimmer Biomet Persona Ti-Nidium Total Knee System
  Interventions: Device: Zimmer Biomet Persona Ti-Nidium Total Knee System

INTERVENTIONS:
Device: Zimmer Biomet Persona Ti-Nidium Total Knee System — Primary Knee Total Arthroplasty

SUMMARY:
The main objectives of this study are to evaluate overall clinical performance and safety of the Persona Ti-Nidium implant in total knee arthroplasty.

DETAILED DESCRIPTION:
The study design is a prospective, multicenter data collection model of the 510(k) cleared Persona Ti-Nidium Total Knee System. The study will require each site to obtain institutional review board (IRB) approval prior to study enrollment. All potential study subjects will be required to participate in the Informed Consent Process.

All study subjects will undergo preoperative clinical evaluations prior to their total knee arthroplasty. Investigators will collect clinical data for a required 10 years. Follow-up clinical visits include Early Post-op, 6 months, 1 year, 2, 3, 5, 7 and 10 years post-operatively.

The objective of this study is to evaluate clinical performance, benefits and safety of the Persona Ti-Nidium implant in total knee arthroplasty.

Specific assessments include:

1. Confirming the long-term safety, performance and clinical benefits of the Persona Ti-Nidium total knee system and instrumentation in primary and revision TKA.
2. Verifying that, under normal use, the performance and clinical benefits of this device and its instrumentation conform to those intended by the manufacturer by recording patient-reported clinical outcomes measures (PROMs) and radiographic outcomes (if available).

ELIGIBILITY:
Inclusion Criteria:

1. Patient is of legal age and skeletally mature
2. Patient is willing and able to provide written Informed Consent by signing and dating the IRB-approved Informed Consent document
3. Patient is willing and able to complete scheduled follow-up evaluations as defined in the study protocol
4. Patient qualifies for total knee arthroplasty based upon physical exam and medical history, and meets the approved indications for use of the Persona Ti-Nidium Knee System and Vivacit-E polyethylene articulating surface
5. Independent of study participation, patient is a candidate for the commercially available Persona Ti-Nidium Knee and Vivacit-E polyethylene articulating surface, implanted in accordance with product labeling

Study Device Inclusion Criteria:

The Persona Ti-Nidium Total Knee is intended for patients with severe pain and disability due to the following:

1. Rheumatoid arthritis, osteoarthritis, traumatic arthritis, polyarthritis.
2. Collagen disorders, and/or avascular necrosis of the femoral condyle.
3. Post-traumatic loss of joint configuration, particularly when there is patellofemoral erosion, dysfunction or prior patellectomy.
4. Moderate valgus, varus, or flexion deformities.

Exclusion Criteria:

1. Patient is unwilling to sign the Informed Consent
2. Patient is currently participating in any other surgical intervention or pain management study
3. Patient is pregnant or considered a member of a protected (vulnerable) population whose inclusion in the study is inappropriate (e.g. prisoner, mentally incompetent)
4. Patient has a mental or neurologic condition who is unwilling or incapable of following postoperative care instructions
5. Patient has a condition which would, in the judgement of the Investigator, place the patient at undue risk or interfere with the conduct of the study
6. Patient is institutionalized or is a known drug abuser, a known alcoholic or cannot understand the requirements of study participation

Study Device Exclusion Criteria

1. Previous history of infection in the affected joint and/or other local/systematic infection that may affect the prosthetic joint
2. Insufficient bone stock on femoral or tibial surfaces
3. Skeletal immaturity
4. Neuropathic arthropathy
5. Osteoporosis or any loss of musculature or neuromuscular disease that compromises the affected limb
6. A stable, painless arthrodesis in a satisfactory functional position
7. Severe instability secondary to the absence of collateral ligament integrity
8. Rheumatoid arthritis (RA) accompanied by an ulcer of the skin or a history of recurrent breakdown of the skin
9. The kinematic alignment surgical technique is contraindicated for patients with greater than 5° valgus deformity with medial collateral ligament (MCL) insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2034-05 (Estimated); Study Completion 2034-05 (Estimated)

PRIMARY OUTCOMES:
Oxford Knee Score (OKS) | 10 years
  A patient reported functional outcome score for knee arthroplasty. This score ranges from 0-48, with higher scores indicating a better outcome.

SECONDARY OUTCOMES:
Knee Society Score (KSS) Expectations (pre and post op) | 10 years
  This is a 3 question form regarding a patient's expectations of the total knee replacement. The pre-op form assesses the patient's expectations of the knee replacement, and the post-op form addresses how the replacement is meeting said expectations. The score ranges from 3-15, with higher scores indicating a better outcome.
EuroQol Five Dimension Five Level (EQ-5D-5L) Outcomes Measure | 10 years
  A questionnaire completed by the patient and assesses his/her general health status. This score ranges from -0.573 to 1, with higher recorded scores indicating better overall health.

CONTACTS AND LOCATIONS:
Overall Officials: Hillary Overholser, Study Director — Zimmer Biomet Assoc Director
Locations (7):
- United States (7):
  - Denver Hip & Knee, Inc., Parker, Colorado
  - MedStar Health Research Institute, Hyattsville, Maryland
  - Mississippi Sports Medicine and Orthopaedic Center, Jackson, Mississippi
  - New Mexico Orthopaedic Associates, Albuquerque, New Mexico
  - Duke University, Durham, North Carolina
  - Rothman Orthopaedic Institute, Philadelphia, Pennsylvania
  - Monument Health Rapid City Hospital, Inc., Rapid City, South Dakota

IPD SHARING:
Plan to Share IPD: No